CLINICAL TRIAL: NCT07272772
Title: Diagnostic Efficacy of 18F-FAPI-74 PET/CT in Patients With Colon Cancer
Brief Title: Colon Cancer Diagnosis With FAPI-PET Imaging
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Colon-FAPI
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-06

CONDITIONS: Colon Cancer
Keywords: Positron Emission Tomography; FAPI; Diagnostics; Imaging; Staging
MeSH Terms: conditions — Colonic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Staging (Experimental): Staging
  Interventions: Device: PET/CT ([F-18]FAPI-74)

INTERVENTIONS:
Device: PET/CT ([F-18]FAPI-74) — PET/CT with FAPI-74 tracer is performed

SUMMARY:
Whole body CT is the primary imaging method in staging and follow-up of colon cancer. Conventional PET-CT with 18F-labeled fluorodeoxyglucose (18F-FDG) has its limitations and has a secondary role in colon cancer protocols. A new PET tracer, fibroblast activation protein inhibitor (FAPI), targeting a protein that is overexpressed by cancer-associated fibroblasts presents a potential new PET imaging tool.

The objective of this prospective study is to evaluate diagnostic efficacy of 18F-FAPI-74 PET/CT in patients with colon cancer. The aim is to evaluate the sensitivity and specificity of 18F-FAPI-74 in detection of local lymph node metastasis and distant metastasis in patient level in patients with colon cancer in primary staging and when suspected recurrence. 100 patients with colon cancer are enrolled and PET/CT studies are performed with the novel 18F-FAPI-74 tracer. The data will be collected between 2024-2026.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary colon cancer with suspicion of mesenteric lymph node metastases in computed tomography before primary cancer operation
* Patients with primary colon cancer with potentially curable metastases
* Patients with suspected metastasis or local recurrence in computed tomography and/or elevated carcinoembryonic antigen (CEA) in cancer surveillance
* WHO performance score 0-2
* Patient signs informed consent form after receiving written information

Exclusion Criteria:

* Vulnerable study subjects such as described in Finnish law clinical studies (disabled, children, pregnant or breast-feeding women, prisoners) will not be included
* Patient is not able to understand purpose of study
* Medical conditions prohibiting whole body PET-CT

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
1) To assess the sensitivity and specificity of 18F-FAPI-74 PET/CT in detection of local lymph node metastasis in patient level in patients with primary colon cancer | 2 years
2) To assess the sensitivity and specificity of 18F-FAPI-74 PET/CT in detection of distant metastasis in patient level in patients with primary colon cancer | 2 years
3) To assess the sensitivity and specificity of 18F-FAPI-74 PET/CT in detection of local lymph metastasis and distant metastasis in patient level in patients with recurrent colon cancer | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Saila Kauhanen, Principal Investigator — Turku PET Centre, Turku University Hospital
Locations (1):
- Turku PET Centre, Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No